CLINICAL TRIAL: NCT06269003
Title: Identifying and Examining the Effects of Source and Presentation on Responses to Electronic Cigarette Public Education Messages in Young Adult Vapers and Non-vapers - Part 2
Brief Title: Responses to Message Source and Presentation Using Psychophysiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Donghee Nicole Lee, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001223; 1K99CA281094-01A1 (NIH)
Record Dates: First submitted 2024-01-17; First posted 2024-02-21 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Expert, one-sided (Experimental): Participants assigned to the expert, one-sidedness condition will receive one-sided e-cigarette messages from an expert source.
  Interventions: Other: Expert, one-sided
- Expert, two-sided (Experimental): Participants assigned to the expert, two-sidedness condition will receive two-sided e-cigarette messages from an expert source.
  Interventions: Other: Expert, two-sided
- Peer, one-sided (Experimental): Participants assigned to the peer, one-sidedness condition will receive one-sided e-cigarette messages from a peer source.
  Interventions: Other: Peer, one-sided
- Peer, two-sided (Experimental): Participants assigned to the peer, two-sidedness condition will receive two-sided e-cigarette messages from a peer source.
  Interventions: Other: Peer, two-sided

INTERVENTIONS:
Other: Expert, one-sided — Participants will view a brief description of an expert source and see one-sided e-cigarette education messages.
  Arms: Expert, one-sided
Other: Expert, two-sided — Participants will view a brief description of an expert source and see two-sided e-cigarette education messages.
  Arms: Expert, two-sided
Other: Peer, one-sided — Participants will view a brief description of a peer source and see one-sided e-cigarette education messages.
  Arms: Peer, one-sided
Other: Peer, two-sided — Participants will view a brief description of a peer source and see two-sided e-cigarette education messages.
  Arms: Peer, two-sided

SUMMARY:
The goal of this clinical trial is to use psychophysiological methods to test the effects of a message source (expert and peer) and message presentation types (one-sided and two-sided) to identify the optimal message type for young adults who vape and do not vape.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-24
* Fluent in English
* Either vaping in the past 30 days or not having vaped in the past 30 days but susceptible to vaping
* Self-reported abstinence of combusted tobacco or marijuana at time of visit

Exclusion Criteria:

* Ages below 18 or above 24
* Not fluent in English
* Not confirmed self-reported abstinence of combusted tobacco or marijuana at time of visit

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donghee N Lee, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Chan Medical School Shaw Building, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on their age (18-24 years old), vaping status (past-30-day vaping and/susceptible to vaping), location (living in the US) between January 2024 to June 2024. The first participant was enrolled in February 18, 2024, and the last participant was enrolled in June 10, 2024.
Groups:
- Expert, One-sided: Participants assigned to the expert, one-sidedness condition were first presented with a brief description of a expert source. They then viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Expert, Two-sided: Participants assigned to the expert, two-sidedness condition were first presented with a brief description of an expert source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
- Peer, One-sided: Participants assigned to the peer, one-sidedness condition were first presented with a brief description of a peer source. They then viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Peer, Two-sided: Participants assigned to the peer, two-sidedness condition were first presented with a brief description of an peer source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
Period: Overall Study
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
Started | 28 | 28 | 28 | 28
Completed | 28 | 28 | 27 (One participant was excluded for being outside the eligible age range.) | 28
Not Completed | 0 | 0 | 1 | 0
Not completed — One participant was excluded for being outside the eligible age range. | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Expert, One-sided: Participants first saw a brief description of a expert source. Then they viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Peer, One-sided: Participants first saw a brief description of a peer source. They then viewed an e-cigarette message that discussed only the health harms of e-cigarette use. This sequence was repeated 18 times during a single study visit.
- Expert, Two-sided: Participants first saw a brief description of an expert source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
- Peer, Two-sided: Participants first saw a brief description of an peer source. They then viewed an e-cigarette message that acknowledged both the potential benefits of e-cigarette use and the associated health risks. This sequence was repeated 18 times during a single study visit.
- Total: Total of all reporting groups
Arm/Group | Expert, One-sided | Peer, One-sided | Expert, Two-sided | Peer, Two-sided | Total
Number analyzed (Participants) | 28 | 27 | 28 | 28 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.25 (1.40) | 21.59 (2.12) | 21.57 (1.75) | 21.82 (1.85) | 21.81 (1.79)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14 | 21 | 17 | 18 | 70
  Male | 11 | 4 | 9 | 6 | 30
  Others | 3 | 2 | 2 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 7 | 3 | 18
  Not Hispanic or Latino | 25 | 22 | 21 | 25 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 4 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 3 | 5
  White | 19 | 17 | 17 | 14 | 67
  More than one race | 2 | 2 | 2 | 1 | 7
  Unknown or Not Reported | 3 | 1 | 4 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 27 | 28 | 28 | 111
Vaping Status [Count of Participants; unit: Participants]
  Current vaping | 15 | 14 | 16 | 16 | 61
  Susceptible to vaping | 13 | 13 | 12 | 12 | 50

OUTCOME MEASURES:

1. Primary Outcome: Visual Attention
Description: Visual attention was assessed by measuring dwell time, which is the length of time participants spent on looking at the specific areas of interest (AOIs) collected in miliseconds. Dwell time values were collected for 18 messages, and aggregated to provide the average dwell time scores for each arm. This was done for each vaping status (current vapers and susceptible non-vapers). Higher dwell time scores indicate higher visual attention, indicating better message outcomes.
Time Frame: The entire duration of message from beginning of its delivery to the completion of viewing, up to 45 minutes.
Population: The data were stratified based on participants' vaping status ("Current vapers" and "Susceptible non-vapers"). The Number of Participants Analyzed for each row reflects the actual number of participants within that vaping status group who were included in the analysis. The Overall Number of Participants Analyzed represents the total number of both subgroups. Any differences have been clarified to specify participant numbers at the row level.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
Number analyzed (Participants) | 28 | 28 | 27 | 28
milliseconds
  Current vapers: number analyzed (Participants) | 15 | 16 | 14 | 16
  Current vapers | 6217.016667 (1278.03706) | 6333.70375 (909.82927) | 6567.725714 (934.62436) | 6667.185625 (633.14744)
  Susceptible non-vapers: number analyzed (Participants) | 13 | 12 | 13 | 12
  Susceptible non-vapers | 6750.67 (798.60759) | 6423.3025 (1069.16916) | 6701.923077 (604.30866) | 6231.6275 (933.71167)

2. Primary Outcome: Allocation of Cognitive Resources
Description: Heart rate values were collected in beats per minute (BPM) on a per-second basis during the presentation of each 18 distinct messages as well as during the immediately preceding black screen (baseline) for each message. Descriptive statistics were used to summarize changes in the BPM values during the message exposure period by comparing the BPM values collected during each message second to the BPM values collected during the immediately preceding baseline period. These change scores were then averaged across all messages within each study arm to generate a mean BPM value per condition, and this was done for each vaping status (current vapers and susceptible non-vapers). Lower BPM values reflect greater cognitive response, therefore indicate better message outcomes.
Time Frame: Baseline and immediately after viewing all the messages (approximately 45 minutes).
Population: n=41 were removed from analysis due to poor quality. The data were stratified based on participants' vaping status ("Current vapers" and "Susceptible non-vapers"). The Number of Participants Analyzed for each row reflects the actual number of participants within that vaping status group who were included in the analysis. The Overall Number of Participants Analyzed represents the total number of both subgroups. Any differences have been clarified to specify participant numbers at the row level.
Measure: Mean (Standard Error); unit: Beats per minute
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
Number analyzed (Participants) | 20 | 18 | 16 | 16
Beats per minute
  Current vapers: number analyzed (Participants) | 9 | 9 | 7 | 7
  Current vapers | -4.885 (1.108) | -4.098 (1.324) | -2.079 (1.239) | -1.652 (1.168)
  Susceptible non-vapers: number analyzed (Participants) | 11 | 9 | 9 | 9
  Susceptible non-vapers | -3.723 (0.834) | -3.444 (0.834) | -3.232 (0.945) | -4.696 (1.119)

3. Primary Outcome: Arousal
Description: Galvanic Skin Response (GSR) values were recorded in microsiemens on a per-second basis during the presentation of each 18 distinct messages as well as during the immediately preceding black screen (baseline) for each message. Descriptive statistics were used to summarize changes in GSR values by comparing each message response to its preceding baseline period. These change scores were then averaged across all messages within each study arm to generate a mean GSR score per condition, and this was done for each vaping status group (current vapers and susceptible non-vapers). Higher GSR values reflect greater physiological arousal, and indicate better message outcomes.
Time Frame: Baseline and immediately after viewing all the messages (approximately 45 minutes).
Population: n=29 were removed from analysis due to poor quality. The data were stratified based on participants' vaping status ("Current vapers" and "Susceptible non-vapers"). The Number of Participants Analyzed for each row reflects the actual number of participants within that vaping status group who were included in the analysis. The Overall Number of Participants Analyzed represents the total number of both subgroups. Any differences have been clarified to specify participant numbers at the row level.
Measure: Mean (Standard Error); unit: microsiemens
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
Number analyzed (Participants) | 21 | 21 | 19 | 21
microsiemens
  Current vapers: number analyzed (Participants) | 9 | 9 | 8 | 9
  Current vapers | 17.225 (272.990) | 597.772 (272.990) | -49.682 (285.129) | 267.135 (272.990)
  Susceptible non-vapers: number analyzed (Participants) | 12 | 12 | 11 | 12
  Susceptible non-vapers | 215.883 (372.223) | -9.867 (372.223) | 526.856 (394.802) | -157.043 (372.223)

4. Secondary Outcome: Attitudes
Description: Participants' self-reported vaping attitudes were measured by using a five-point bipolar scale using 7 subscale items assessing whether participants thought vaping was enjoyable, healthy, safe, fun, smart, cool, and attractive on a scale from 1 (negative attitudes) to 5 (positive attitudes). Items were summed and averaged to create a single composite score, and this was done for each arm for each vaping status. Higher scores indicate more positive e-cigarette attitudes, therefore worse outcomes.
Time Frame: After exposure to all messages, approximately up to 45 minutes.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
Number analyzed (Participants) | 28 | 28 | 27 | 28
score on a scale
  Current vapers: number analyzed (Participants) | 15 | 16 | 14 | 16
  Current vapers | 1.9619 (.45326) | 2.1771 (.54931) | 2.1480 (.62299) | 1.8824 (.39817)
  Susceptible non-vapers: number analyzed (Participants) | 13 | 12 | 13 | 12
  Susceptible non-vapers | 1.6593 (.40632) | 1.5833 (.48141) | 1.6044 (.51228) | 1.8571 (.40913)

5. Secondary Outcome: Behavioral Intentions
Description: Participants' vaping intentions was measured by using a 3 subscale items assessing participants' intentions to vape: soon/anytime during the next year/would use offered by one of their best friends, on a scale from 1 (Definitely not) to 5 (Definitely yes). Items were summed and averaged to create a single composite score. This was done for each vaping status (current vapers and susceptible non-vapers). Higher scores indicate greater vaping intentions, therefore indicating worse outcome.
Time Frame: After exposure to all messages, approximately up to 45 minutes.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Expert, One-sided | Expert, Two-sided | Peer, One-sided | Peer, Two-sided
Number analyzed (Participants) | 28 | 28 | 27 | 28
score on a scale
  Current vapers: number analyzed (Participants) | 15 | 16 | 14 | 16
  Current vapers | 2.7556 (0.98776) | 3.0313 (0.87817) | 3.0238 (0.90075) | 2.5833 (0.96992)
  Susceptible non-vapers: number analyzed (Participants) | 13 | 12 | 13 | 12
  Susceptible non-vapers | 1.3333 (.49065) | 1.0278 (.09623) | 1.2564 (.47442) | 1.3056 (.30011)

ADVERSE EVENTS:
Time Frame: Each adverse event or serious adverse event was monitored and assessed throughout the entire duration of the participant's lab visit, from the moment a participant showed up to the lab until the study completed, which lasted approximately 1 hour per participant.
Description: The study used a non-systematic assessment method, where adverse events were monitored through participants' verbal reports and observing participants' behaviors. No adverse events were reported by participants or observed during the study duration.
Groups:
- Expert 1-sided: During the reporting period, no adverse events were observed or reported among participants in the expert 1-sided arm.
  All 28 participants completed the study phase without any clinical complaints, side effects, or complications attributed to the intervention.
- Expert 2-sided: During the reporting period, no adverse events were observed or reported among participants in the expert 2-sided arm.
  All 28 participants completed the study phase without any clinical complaints, side effects, or complications attributed to the intervention.
- Peer 1-sided: During the reporting period, no adverse events were observed or reported among participants in the peer 1-sided arm.
  All 27 participants completed the study phase without any clinical complaints, side effects, or complications attributed to the intervention.
- Peer 2-sided: During the reporting period, no adverse events were observed or reported among participants in the peer 2-sided arm.
  All 28 participants completed the study phase without any clinical complaints, side effects, or complications attributed to the intervention.
Arm/Group | Expert 1-sided | Expert 2-sided | Peer 1-sided | Peer 2-sided
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT06269003/Prot_001.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT06269003/SAP_000.pdf